CLINICAL TRIAL: NCT03492775
Title: Prospective Randomized Evaluation of Single Agent GA101 Versus GA101 Plus Bendamustine Followed by GA101
Brief Title: First Line Therapy of Advanced Stage Follicular Lymphoma in Patients < 60 Years Not Eligible fo Standard Immunochemotherapy and in All Patients ≥ 60 Years
Acronym: GABe2016
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Wolfgang Hiddemann (Other)
Collaborators: Hoffmann-La Roche (Industry); Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Wolfgang Hiddemann, Prof. Dr. med. Wolfgang Hiddemann, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000755-27
Record Dates: First submitted 2017-12-04; First posted 2018-04-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Indolent Non-hodgkin Lymphoma
Keywords: indolent lymphoma; Obinutuzumab; GA101; Bendamustine; medically non-fit patients
MeSH Terms: interventions — obinutuzumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A:Obinutuzumab single agent (Active Comparator): Obinutuzumab flat dose of 1000 mg on Day 1 of each of four 28 -day cycles and on Days 8 and 15 of Cycle 1
  If at least 'stable disease':
  Obinutuzumab flat dose of 1000 mg at weeks 21, 29, 37 and 45
  Interventions: Drug: Obinutuzumab
- Arm B:Obinutuzumab plus Bendamustine (Active Comparator): Obinutuzumab flat dose of 1000 mg on Day 1 of each of four 28 -day cycles and on Days 8 and 15 of Cycle 1 plus Bendamustine 70 mg/m2 iv d1+2 of each of four 28 -day cycles
  If at least 'stable disease':
  Obinutuzumab flat dose of 1000 mg at weeks 21, 29, 37 and 45
  Interventions: Drug: Obinutuzumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab (GA 101) is a first-in-class, potent, intravenously administered type II anti-CD 20 antibody that is developed by Roche AG for the treatment of B-cell malignancies.
  Other Names: GA 101
Drug: Bendamustine — Bendamustine belongs formally to the alkylators, but has been shown to have a unique mechanism of action. The dose limiting toxicity of bendamustine is its reversible suppression of bone marrow function with drops in leukocyte and thromobocyte counts.
  Other Names: Bendamustine hydrochloride; Ribomustin
  Arms: Arm B:Obinutuzumab plus Bendamustine

SUMMARY:
The objective of this study is to test the efficacy and toxicity of a combined OBINUTUZUMAB/bendamustine therapy or single agent OBINUTUZUMAB in younger (< 60 years) medically non-fit, 'compromised' patients and in all older patients (≥ 60 years). For the assessment of the antilymphoma activity the overall response rate (ORR)" will be applied as primary endpoint.

Overall response is defined as complete or partial response after 19 - 21 weeks.

DETAILED DESCRIPTION:
Study design:

This is a randomized, open-label, multicenter phase II trial with a parallel-group design of two groups.

Randomization and Interventions:

Randomization between Obinutuzumab single agent treatment versus Obinutuzumab plus Bendamustine followed by Obinutuzumab

Treatment plans:

Arm A: Obinutuzumab single agent Obinutuzumab flat dose of 1000 mg on Day 1 of each of four 28 -day cycles and on Days 8 and 15 of Cycle 1

If at least 'stable disease':

Obinutuzumab flat dose of 1000 mg at weeks 21, 29, 37 and 45 Arm B: Obinutuzumab plus Bendamustine Obinutuzumab flat dose of 1000 mg on Day 1 of each of four 28 -day cycles and on Days 8 and 15 of Cycle 1 plus Bendamustine 70 mg/m2 iv d1+2 of each of four 28 -day cycles

If at least 'stable disease':

Obinutuzumab flat dose of 1000 mg at weeks 21, 29, 37 and 45

The project attempts to establish an evidence based treatment strategy for medically non-fit advanced stage FL-patients who are not eligible for standard therapeutic immunochemotherapy approaches to improve their long term perspectives.

It will furthermore provide a prospectively generated data set which will link performance in the assessment scores IADL, G8 and CIRS-G to medical fitness as judged by the treating physician. The generated data will allow using geriatric and functional tests to define medical fitness and to provide a more solid basis for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Medically nonfit" patients < 60 years defined by

  o ECOG > 2 or ECOG 0-2 with co-morbidities excluding intensive therapy according to local investigator's discretion
* All patients ≥ 60 years in case of decision of investigator and patient to apply a reduced Treatment
* Documentation of the CIRS-G, IADL, G8 and ECOG Scores before start of treatment
* Histologically confirmed follicular lymphoma grade I, II or IIIa with material available for central pathology review
* Stage III/IV or stage II without the option of curative radiotherapy
* Age > 18 years
* No prior therapy
* Presence of at least one of the following symptoms or conditions requiring initiation of treatment:

  * Bulky disease according to the GELF criteria: nodal or extranodal mass > 7cm in its greater diameter
  * B symptoms (fever, drenching night sweats, or unintentional weight loss of >10% of normal body weight over a period of 6 months or less)
  * Hematopoietic insufficiency (at least one of the following: granulocytopenia <1500 cells/μl, Hb < 10 g/dl, thrombocytopenia <100.000 cells/μl)
  * Compressive syndrome
  * Pleural/peritoneal effusion
  * Symptomatic nodal or extranodal manifestations
* At least one bi-dimensionally measurable lesion (> 1.5 cm in its largest dimension by CT scan or MRI)
* Adequate hematologic function (unless abnormalities are related to NHL), defined as follows:

  * hemoglobin ≥ 9.0 g/dl
  * absolute neutrophil count ≥ 1500 /μL
  * platelet count ≥ 75000 /μl
* Women who are not breast feeding, are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and during the 18 months thereafter.
* Men who agree not to father a child during participation in the trial and during the 18 months thereafter.
* Written informed consent form

Exclusion Criteria:

"Medically fit" patients < 60 years with the option for more intensive induction therapy such as R-CHOP

* Transformation to high-grade lymphoma (secondary to "low-grade" follicular lymphoma)
* Grade IIIb follicular lymphoma
* Presence or history of CNS disease (either CNS lymphoma or lymphomatous meningitis).
* Regular use of corticosteroids during the last 4 weeks, unless administered at a dose equivalent to < 20 mg/day prednisone.
* Prior (< 3 years) or concomitant malignancies except non-melanoma skin cancer or adequately treated in situ cervical cancer.
* Major surgery (excluding lymph node biopsy) within 28 days prior to registration.
* Necessity of rapid cytoreduction
* Serious underlying medical conditions, which could impair the ability of the patient to tolerate the therapy offered in this trial (e.g. ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease).
* Severe hepatic impairment (serum bilirubin > 3.0 mg/dl)
* Known sensitivity or allergy to murine products
* Known hypersensitivity to any of the study drugs
* Treatment within a clinical lymphoma trial within 30 days prior to trial entry
* Positive test results for chronic HBV infection (defined as positive HBsAg serology) (mandatory testing) Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable, provided that they are willing to undergo monthly DNA testing. Patients who have protective titers of hepatitis B surface antibody (HBSAb) after vaccination or prior but cured hepatitis B are eligible.
* Positive test results for hepatitis C (mandatory hepatitis C virus [HCV] antibody serology testing). Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA
* Known history of HIV seropositive status.
* Patients with a history of confirmed PML
* Vaccination with a live vaccine within 28 days prior to registration
* Prior organ, bone marrow or peripheral blood stem cell transplantation
* Any other co-existing medical or psychological condition that will preclude participation in the study or compromise the ability to understand its nature,meaning and implications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ORR | week 19 to 21
  Overall response is defined as complete or partial response at the end of the initial treatment phase (after 19-21 weeks).

SECONDARY OUTCOMES:
Event free survival, EFS | through study completion, up to 5 years
  Response in accordance with the 2007 Revised Response Criteria for the time from the day of randomization to the date of first documented disease progression, death by any cause, or institution of a new anti-lymphoma treatment.
CR | End of Induction of each patient, week 19 - 21
  Rate of patients who has a complete response (CR) at the end of induction randomization
TTF | Through study completion, up to 5 years
  The time to treatment failure will be measured from the day of randomization to the date of failure of initial treatment (no response) or first documented disease progression or death by any cause.
PFS | Through study completion, up to 5 years
  progression-free survival will be measured from the day of randomization to the date of first documented disease progression or death by any cause.
RD | week 19 up to 5,5 years follow up
  Duration of remission will be measured for responding patients from the end of initial treatment to the date of first documented disease progression or death by any cause.
Time to next anti-lymphoma treatment | Through study completion, up to 6.5 years
  will be measured from the date of randomization to the date of first documented start of a new chemotherapy, radiotherapy or immunotherapy.
Overall Survival | Through study completion, up to 5 years
  will be determined from the date of randomization to the date of death irrespective of cause.
Number of SAEs | Through study completion, up to 5 years
  Therapy-related toxicities according to the NCI-CTC-criteria will be compared for both treatment arms during the initial treatment and the consolidation treatment period.
Frequency of Hospitalization | Through study completion, up to 3 years (per patient)
  The days of hospitalisation will be compared for both treatment arms during the initial treatment, the consolidation treatment period and the first two years after the end of consolidation.
Duration of Hospitalization | Through study completion, up to 3 years (per patient)
  The duration of hospitalisation will be compared for both treatment arms during the initial treatment, the consolidation treatment period and the first two years after the end of consolidation.
Supportive Care | Through study completion, up to 5 years
  The number of blood transfusions, the application of growth factors and the days of treatment with i.v. antibiotics will be compared for both treatment arms
Incidence of secondary transformation to aggressive lymphoma | Through study completion, up to 5 years
  Incidence of secondary transformation to aggressive lymphoma
Number of AEs | Through study completion, up to 5 years
  Incidence of secondary malignancies
Number of participants that had completed the therapy regularly (including: Total cumulative dose of obinutuzumab and bendamustine, number of cycles, duration of treatment) | Through study completion, up to 5 years
QoL | Through study completion, up to 5 years
  Quality of Life Analysis scale measurements using the QLQ-C30 questionnaires are collected over time and will be compared for patients receiving OBINUTUZUMAB single agent versus OBINUTUZUMAB plus bendamustine.
Comorbidity assessment will be performed by using the Instrumental Activities of Daily Living (=IADL) | Through study completion, up to 6.5 years
  With the Instrumental Activities of Daily Living (=IADL) the functional status) will be analysed (=instrument to assess independent living skills) The instrument is most useful for identifying how a person is functioning at the present time and for identifying improvement or deterioration over time. There are 8 domains of function measured with the Lawton IADL scale. Historically, women were scored on all 8 areas of function; men were not scored in the domains of food preparation, housekeeping, laundering. However, current recommendations are to assess all domains for both genders. Persons are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
Comorbidity assessment will be performed by using the Cumulative Illness Rating Scale for Geriatrics (CIRS-G) | Through study completion, up to 5 years
  This can be used to measure the burden of current and chronic illnesses in the older adult.This scoring system measures the chronic medical illness ("morbidity") burden while taking into consideration the severity of chronic diseases in 14 items representing individual body systems.
  The general rules for severity rating are:
  0→No problem affecting that system.
  1. Current mild problem or past significant problem.
  2. Moderate disability or morbidity and/or requires first line therapy.
  3. Severe problem and/or constant and significant disability and/or hard to control chronic problems.
  4. Extremely severe problem and/or immediate treatment required and/or organ failure and/or severe functional impairment.
Comorbidity assessment will be performed by using the G 8 (=geriatric) 8 screening score | Through study completion, up to 5 years
  The G8 screening tool was developed to separate fit older cancer patients who were able to receive standard treatment from those that should undergo a geriatric assessment to guide tailoring of therapy. The assessment includes (instrumental) activities of daily living, cognition, mood, nutritional status, mobility, polypharmacy and social support. G8 is an independent predictor of mortality within the first year after inclusion (hazard ratio 3.93; 95 % confidence interval 1.67-9.22, p < 0.001). The G-8 Score is a screening tool containing 8 questions. The total G-8 score lies between 0 and 17. A higher score indicates a better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hiddemann, Prof.Dr., Study Chair — Hospital of the University of Munich
Locations (1):
- Klinikum der Universität München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No